CLINICAL TRIAL: NCT00649792
Title: Phase 3 Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR in Patients With Multiple Sclerosis Who Participated in the MS-F204 Trial
Brief Title: Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR in Patients With Multiple Sclerosis Who Participated in the MS-F204 Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-F204 EXT
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MS; walking; leg strength; demyelination
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fampridine-SR — Tablets, 10 mg, BID (twice daily)
  Other Names: 4-aminopyridine

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and activity of Fampridine-SR when administered for up to 36 additional months in patients who previously participated in the MS-F204 study or until it becomes commercially available, whichever comes first.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result, patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR is an experimental drug that has been reported to possibly improve muscle strength and walking ability for some people with MS. This study will evaluate the effects and possible risks of taking Fampridine-SR in MS patients over a long period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been previously enrolled in the Acorda Therapeutics MS-F204 study and received either Fampridine-SR or placebo
* Patient with clinically defined multiple sclerosis (the diagnostic criteria based on: McDonald WI, et al. Recommended Diagnostic Criteria for Multiple Sclerosis: Guidelines from the International Panel on the Diagnosis of Multiple Sclerosis. Annals of Neurology. 2001; 50: 121-127)
* Patient must be at least 18 years of age. Any patient who is now over the age of 70 must be in good overall health in the judgment of the investigator
* Patient must be of adequate cognitive function, as judged by the Investigator
* Patients who are women of childbearing potential must have a negative urine pregnancy test at the screening visit

Exclusion Criteria:

* Female patients who are either pregnant or breastfeeding.
* Women of childbearing potential who are not using a specified birth control method
* Patients discontinued prematurely from the MS-F204 study
* Patients with a history of seizures or with evidence of past, or possible epileptiform activity on an EEG
* Patient with either a clinically significant abnormal ECG or laboratory values at the MS-F204 EXT screening visit
* Patient with severe renal impairment
* Patient with angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality, as judged by the Investigator
* Patient with a known allergy to pyridine-containing substances or any of the inactive ingredients of the Fampridine-SR tablet
* Patient who has received an investigational drug (other than Fampridine-SR or placebo under MS-F204 study) within 30 days of the MS-F204EXT screening visit or a patient who is scheduled to enroll in an investigational drug trial at any time during this study
* Patient who has a history of drug or alcohol abuse within the past year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Faust, Study Director — Acorda Therapeutics
Locations (42):
- United States (38):
  - Barrow Neurology Clinic, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Neurological Associates, Fayetteville, Arkansas
  - Alta Bates Summit Medical Center - Research and Education Institute, Berkeley, California
  - USC, Keck School of Medicine Health Care Consultation Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - Yale University MS Center, New Haven, Connecticut
  - Shepherd Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Consultants in Neurology, Ltd., Northbrook, Illinois
  - Indiana University MS Center, Indianapolis, Indiana
  - Associates in Neurology, PSC, Lexington, Kentucky
  - Maryland Center for MS, Baltimore, Maryland
  - Lahey Clinic, Lexington, Massachusetts
  - Wayne State University, Department of Neurology, Detroit, Michigan
  - The Schapiro Center for MS, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - UMDNJ, Newark, New Jersey
  - Gimbel MS Center at Holy Name Hospital, Teaneck, New Jersey
  - Jacobs Neurological Institute Buffalo General Hospital, Buffalo, New York
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - Columbia University Multiple Sclerosis Clinical Care Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - CMC - Neuroscience & Spine Institute, Division of Neurology, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University, Dept of Neurology, M.S. Research, Winston-Salem, North Carolina
  - The Center for Neurological Services, Bismarck, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University MS Center, Columbus, Ohio
  - Oregon Health & Science University, MS Center of Oregon, UHS-42, Portland, Oregon
  - Thomas Jefferson University Physicians, Philadelphia, Pennsylvania
  - Neurological Research Center, Inc., Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - MS Center at Evergreen, Kirkland, Washington
  - CAMC Health Education & Research Institute, Charleston, West Virginia
  - Center for Neurological Disorders of Aurora, St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - University of British Columbia, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - River Valley Health c/o Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QEII Health Sciences Centre, Nova Scotia Rehabilitation Centre Site, Halifax, Nova Scotia

REFERENCES:
- See also: Click here for more information about Fampridine-SR clinical trials — http://www.acorda.com/clinical.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Fampridine-SR: Tablets, 10 mg, BID
Period: Overall Study
Arm/Group | Fampridine-SR
Started | 214
Completed | 146
Not Completed | 68

BASELINE CHARACTERISTICS:
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 201
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 201
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Secondary Outcome: Timed 25-Foot Walk (T25FW)
Time Frame: Week 2, 14, 26, continuing every 26 weeks until the Final Visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: feet/seconds
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 211
feet/seconds
  (N=209) >0-8 Weeks | 2.60 (0.86)
  (N=197) >8-16 Weeks | 2.53 (0.93)
  (N=201) >16-42 Weeks | 2.52 (0.96)
  (N=172) >42-68 Weeks | 2.46 (1.02)
  (N=160) >68-94 Weeks | 2.37 (1.04)
  (N=151) >94-120 Weeks | 2.35 (1.10)
  (N=143) >120-146 Weeks | 2.27 (1.06)
  (N=33) >146-172 Weeks | 2.17 (1.07)
  (N=2) >172-198 Weeks | 1.85 (0.56)

2. Secondary Outcome: Subject Global Impression (SGI)
Description: For the SGI, the potential responses to the effects of the investigational drug during the preceding week were 1=terrible, 2=unhappy, 3=mostly dissatisfied, 4=neutral/ mixed, 5=mostly satisfied, 6=pleased, and 7=delighted.
Time Frame: Visit 1 and every clinic visit thereafter (other than the follow-up visit)
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: 1-7 scale rating
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 214
1-7 scale rating
  (N=214) >0-8 Weeks | 4.67 (1.15)
  (N=200) >8-16 Weeks | 4.70 (1.28)
  (N=199) >16-42 Weeks | 4.77 (1.29)
  (N=183) >42-68 Weeks | 5.04 (1.19)
  (N=173) >68-94 Weeks | 4.95 (1.20)
  (N=167) >94-120 Weeks | 4.97 (1.27)
  (N=153) >120-146 Weeks | 5.15 (1.11)
  (N=35) >146-172 Weeks | 4.94 (1.39)
  (N=2) >172-198 Weeks | 5.50 (0.71)

3. Secondary Outcome: Clinician's Global Impression (CGI)
Description: The potential responses were 1=very much improved, 2=much improved, 3=somewhat improved, 4=no change, 5=somewhat worse, 6=much worse, and 7=very much worse.
Time Frame: Visit 1 and every clinic visit thereafter
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: 1-7 scale rating
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 213
1-7 scale rating
  (N=213) >0-8 Weeks | 3.38 (0.84)
  (N=202) >8-16 Weeks | 3.27 (0.90)
  (N=208) >16-42 Weeks | 3.48 (0.98)
  (N=181) >42-68 Weeks | 3.42 (0.92)
  (N=172) >68-94 Weeks | 3.58 (1.14)
  (N=168) >94-120 Weeks | 3.66 (1.19)
  (N=154) >120-146 Weeks | 3.65 (1.16)
  (N=35) >146-172 Weeks | 3.96 (1.17)
  (N=2) >172-198 Weeks | 2.50 (0.71)

4. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: The EDSS was used to grade patient disability on a scale from 0.0 (normal neurological exam) to 10.0 (death)
Time Frame: The Screening Visit, Visit 6, Final Visit or Early Termination Visit (if applicable)
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: 0-10 rating scale
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 213
0-10 rating scale
  (N=213) Baseline | 5.64 (1.11)
  (N=163) >94-120 Weeks | 5.86 (1.05)

5. Primary Outcome: Summary of Treatment Emergent Adverse Events (TEAE).
Description: All adverse events reported were treatment emergent. Therefore, events that had a date of onset, or worsening, on or after the start of the open-label drug and up to 14 days after the last dose (for non-serious events) or up to 30 days after the last dose (for SAEs) were summarized. Any abnormal clinically significant changes in physical examination, medical history, clinical laboratory testing, 12-lead ECG, and standard EEG testing were captured as adverse events.
Time Frame: up to 40 months
Population: Safety Population. No imputation for missing data
Measure: Number; unit: participants
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 214
participants
  Patients with Any TEAE | 205
  Patients with Any Serious TEAE | 39
  Patients with Any Treatment-Related AE | 46
  Patients Withdrawn due to AE | 7
  Patients who Died | 1
  Maximum Severity/Paitents with Any TEAE - Mild | 29
  Maximum Severity/Patients with Any TEAE - Moderate | 120
  Maximum Severity/Patients with Any TEAE - Severe | 56

ADVERSE EVENTS:
Arm/Group | Fampridine-SR
Serious Adverse Events (participants affected / at risk) | 39/214
Other Adverse Events (participants affected / at risk) | 205/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR (N=214)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1)
Arthritis Infective (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Clostridium Colitis (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Device Related Infection (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Puncture Headache (Injury, poisoning and procedural complications) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 5 (6)
Muscle Spasticity (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Orbital Infection (Infections and infestations) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1)
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR (N=214)
Adverse Drug Reaction (General disorders) | 18 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (43)
Asthenia (General disorders) | 12 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 23 (30)
Balance Disorder (Nervous system disorders) | 23 (29)
Blood Creatine Phosphokinase Increased (Investigations) | 13 (15)
Contusion (Injury, poisoning and procedural complications) | 30 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Depression (Psychiatric disorders) | 14 (19)
Dizziness (Nervous system disorders) | 24 (30)
Fall (Injury, poisoning and procedural complications) | 88 (182)
Fatique (General disorders) | 37 (39)
Headache (Nervous system disorders) | 15 (21)
Hypoaesthesia (Nervous system disorders) | 13 (13)
Influenza (Infections and infestations) | 15 (17)
Insomnia (Psychiatric disorders) | 16 (18)
Multiple Sclerosis Relapse (Nervous system disorders) | 61 (102)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 (14)
Muscle Spasticity (Nervous system disorders) | 29 (33)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 38 (48)
Nasopharyngitis (Infections and infestations) | 21 (25)
Nausea (Gastrointestinal disorders) | 27 (33)
Oedema Peripheral (General disorders) | 37 (43)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 29 (37)
Pyrexia (General disorders) | 12 (15)
Rash (Skin and subcutaneous tissue disorders) | 12 (13)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 13 (14)
Sinusitis (Infections and infestations) | 11 (12)
Skin Laceration (Injury, poisoning and procedural complications) | 12 (13)
Upper Respiratory Tract Infection (Infections and infestations) | 31 (39)
Urinary Tract Infection (Infections and infestations) | 75 (148)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.